CLINICAL TRIAL: NCT03315858
Title: NFAT (Nuclear Factor of Activated T-cells)-Regulated Gene Expression After Tacrolimus -the Basis for Future Tailored Immunosuppression-
Brief Title: NFAT-regulated Gene Expression After Tacrolimus
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: NFAT1
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: NFAT Regulated Gene Expression in Tacrolimus Treated Patients
Keywords: NFAT; gene expression; tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study is measurement of NFAT-RGE (IL-2 (interleukin-2), IFN-γ (interferon-gamma), GM-CSF (granulocyte monocyte colony stimulating factor)) after tacrolimus (TAC) in de-novo immunosuppressed patients after liver transplantation (LT), to test the hypothesis that in de-novo TAC patients receiving mycophenolate mofetil (MMF) and steroids after LT there is an inverse correlation of NFAT-RGE and TAC peak levels at 1.5 hours after TAC intake.

DETAILED DESCRIPTION:
The trial will be conducted as a prospective, longitudinal study. The study is a single-centre study performed at the Medical University of Graz, Department of Surgery, Division of Transplant Surgery and the Department of Blood Group Serology and Transfusion Medicine, Medical University of Graz.

All the patients on the LT wailting list at the Division of Transplant Surgery, Medical University of Graz are screened according to both inclusion and exclusion criteria. The study period is 1 year. One NFAT-RGE baseline measurement is performed directly before LT; NFAT-RGE-measurements after LT are performed at clearly defined timepoints.

Study population. As a pilot trial this study comprises of 15 patients who will undergo LT

Objectives:

* To test the hypothesis that in de-novo TAC patients receiving mycophenolate mofetil (MMF) and steroids after LT there is an inverse correlation of NFAT-RGE and TAC peak levels at 1.5 hours after TAC intake
* To correlate both NFAT-RGE and TAC (trough and peak) levels with rejection episodes and TAC side effects

Approach:

NFAT-RGE is determined in 15 patients just before LT, and after LT after 1 day, 1 week, 2 weeks, and after 1, 6 and 12 months.

Methods. Heparinized peripheral blood is stimulated with 1 ml of complete Roswell Park Memorial Institute (RPMI) 1640 medium containing 100 ng/ml phorbol 12-myristate 13-acetate (PMA) and 5 mcg/ml ionomycin (Sigma-Aldrich Corp., St.Louis, MO, USA) for 3 hours at 37°C. Following ex vivo immune activation, after red cell lysis with ACK buffer (0.15 M NH4CL, 1.0 mM KHCO3), leukocytes are lysed with 400 mcl of MagNA-Pure lysis buffer supplemented with an additional 1% (W/v) of dithiothritol (RAS, Mannheim, Germany), and the sample is frozen at -70°C. After thawing, mRNA is isolated with the RNA Blood mini Kit (Quiagen) device using the mRNA standard protocol for cells. RNA is reverse transcribed using SuperScript III First-Strand Synthesis System for RT-PCR (Invitrogen, life technologies). The 3 NFAT-regulated genes (IFN-γ, IL-2, GM-CSF) were identified as suitable genes for this essay from previous studies [18, 26]. Target mRNA sequences of IFN- γ, IL-2, GM-CSF and 3 reference genes are amplified using commercially available PrimePCR ddPCR Gene Expression Probe Assays (Biorad) by digital PCR (Biorad).

The RGE after TAC intake is calculated as cpeak/c0x100, where c0 is the adjusted number of transcripts at the TAC predose level and cpeak is the number of transcripts 1.5 (c1.5) hours after drug intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Liver transplantation
* Informed consent

Exclusion Criteria:

* Patients < 18 of years
* Patients taking actively part in a different interventional trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As a pilot trial this study comprises of 15 patients who will undergo liver transplantation.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
correlation of NFAT-RGE and TAC peak levels | 1 year
  Calculation: cpeak/c0x100

SECONDARY OUTCOMES:
correlation of both NFAT-RGE and TAC (trough and peak) levels with rejection episodes and TAC side effects | 1 year
  Calculation: cpeak/c0x100

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Klin. Abteilung für Transplantationschirurgie, Graz, Austria